CLINICAL TRIAL: NCT04226222
Title: Bringing Semi-quantitative PET-TDM FDG Data and Texture Analysis to Clinical, Histological and Immuno-histochemical Characteristics of Primary Mammary Tumors Triple Negatives
Brief Title: Bringing of PET-TDM FDG in the Determination of the Characteristics of Primary Mammary Tumors TrIple Negatives
Acronym: FICTION
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Institut Cancerologie de l'Ouest (Other)
Responsible Party: Sponsor
Other Study IDs: ICO-2019-03
Record Dates: First submitted 2020-01-09; First posted 2020-01-13 (Actual); Last update posted 2023-02-21 (Actual); Status verified 2022-08

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Triple negative Breast Cancer: Triple Negative Breast Cancer operatable from the outset
  Interventions: Diagnostic Test: TEP-TDM FDG

INTERVENTIONS:
Diagnostic Test: TEP-TDM FDG — Semi-quantitative PET-TDM FDG Data and Texture Analysis

SUMMARY:
"Triple Negative" breast cancers are a heterogeneous group characterized by the absence of hormone receptors to estrogen, progesterone and the absence of expression or amplification of the HER-2 gene. This type of cancer is associated with an adverse clinical profile with a high risk of early metastatic relapse. Accurate identification of prognostic factors, as well as predictors of therapeutic response, and the contribution of targeted therapies are avenues for improving the management and survival of patients with these cancers. Such an approach requires optimal biological characterization, allowing us to understand the complexity of this group of tumors, and requires multidisciplinary collaboration in clinical trials involving anatomopathology, oncology and morpho-functional imaging.

The investigator's goal is to characterize by innovative methods (anatomo-pathological in particular Of Immunohistochemistry, and morpho-functional imaging (TEP-TDM FDG) semi-quantitative and texture) in a population of Triple Negative Breast Cancer scans better knowledge of this entity that can lead to the development of relevant therapeutic strategies and especially more adapted in the context of precision and personalized medicine.

DETAILED DESCRIPTION:
120 consecutive patients with "Triple Negative" breast cancers operatable from the outset will be included in the study

* To assess the prognostic value of the texture parameters of PET-TDM FDG on event-free survival at 2 years.
* To assess the prognostic value of standard parameters (clinical, standard histology, conventional imaging), semi-quantitative PET-TDM FDG and innovative Immuno-histochemistry parameters for 2-year event-free survival .
* To assess correlations between continuous PET-TDM FDG texture parameters and Immuno-histochemistry.
* To assess the multivariate prognostic value of standard parameters, PET-TDM FDG imaging parameters and Immuno-histochemistry defined as relevant to 2-year event-free survival .
* Construction of an optimal prognostic nomogram combining independent parameters to isolate different prognostic subgroups.

ELIGIBILITY:
Inclusion Criteria:

* Patient with biopsy-proven triple-negative breast cancer, newly diagnosed, naïve from any treatment.
* Age - 18.
* Performance Status (PS) : 0 or 1.
* No metastasis on the extension balance.
* Treatment provided immediately by lumpectomy or mastectomy, and accepted by the patient.

Exclusion Criteria:

* Severe illness or comorbidity at risk.
* A history of cancer within 5 years, with the exception of skin carcinomas (other than melanoma) or in-situ cervical carcinomas.
* Patient candidate for neo-adjuvant therapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients with triple negative breast cancer operatable from the outset will be
Sampling Method: Non-Probability Sample
Enrollment: 132 (Actual)
Dates: Start 2019-11-05 (Actual); Primary Completion 2022-10-22 (Actual); Study Completion 2024-10-22 (Estimated)

PRIMARY OUTCOMES:
Assess the prognostic value of the texture parameters of PET-TDM FDG on event-free survival at 2 years. | 2 years
  The 2-year event-free survival rate based on the texture parameters of the PET-TDM FDG.
  Event free survival is the duration between the date of diagnosis and the date of the first event (relapse, death) or the date of the last news without event.

SECONDARY OUTCOMES:
assess the prognostic value of standard parameters (clinical, standard histology, conventional imaging), semi-quantitative PET-TDM FDG and innovative Immunohistochemistry parameters for 2-year event-free survival . | 2 years
  2-year event-free survival rate based on univariate analysis of standard, semi-quantitative parameters of PET-TDM FDG and innovative Immunohistochemistry parameters.
To assess the correlations between continuous texture parameters in PET-TDM FDG and Immunohistochemistry. | 2 years
  Correlation coefficients between the continuous criteria of the FDG PET texture parameters and those of the Immunohistochemistry.
assess the multivariate prognostic value of standard parameters, PET-TDM FDG imaging parameters and Immunohistochemistry defined as relevant to 2-year event-free survival | 2 years
  2-year event-free survival rate in multivariate analysis according to standard parameters, PET-TDM FDG imaging parameters and Immunohistochemistry.
Construction of an optimal prognostic nomogram combining independent parameters to isolate different prognostic subgroups | 2 years
  2-year event-free survival rate depending on the risk groups determined from the nomogram score.

CONTACTS AND LOCATIONS:
Overall Officials: Caroline ROUSSEAU, MD, PhD, Principal Investigator — caroline.rousseau@ico.unicancer.fr
Locations (2):
- France (2):
  - Institut de Cancérologie de l'Ouest, Angers
  - Institut de Cancerologie de L'Ouest, Saint-Herblain